CLINICAL TRIAL: NCT03515746
Title: 3D or 2D Upper Extremity Exergaming for Persons With Parkinson's Disease
Acronym: 10Cubes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Collaborators: European Regional Development Fund (Other); Slovenian Research Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URIS201801
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Parkinson Disease
Keywords: exergaming; physiotherapy; upper extremities; telerehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergaming2D (Active Comparator): The participants will practise grab and grasp through exergaming in virtual environment (VE) on a laptop computer. During the task, they will sit in a comfortable chair in front of the screen.
  Interventions: Device: Exergaming in virtual environment
- Exergaming3D (Active Comparator): The participants will practise grab and grasp through exergaming in virtual environment (VE) in 3D VE using Oculus Rift CV1 3D goggles. During the task, they will sit in a comfortable chair with head-mounted 3D display.
  Interventions: Device: Exergaming in virtual environment

INTERVENTIONS:
Device: Exergaming in virtual environment — The "10 cubes" task will be performed in virtual environment - either in 2D on a laptop computer or in 3D using 3D goggles

SUMMARY:
A pilot study with the "10cubes" for small and precise movements and training in the virtual environment will be carried out. We will recruit at least 20 persons with Parkinson's disease to participate in the study. Such activities can increase participation, slow down the progress of the disease and contribute to the functional improvements of the hand that lead to the increased quality of life. The movement of the hand will be assessed with a small 3D camera, also suitable for the estimation of kinematic parameters. Participants will be randomized into 2 groups; one group using an LCD screen and the other using 3D goggles (Oculus Rift CV1) enabling them to carry out the task in virtual environment. Both groups will take 10 training sessions within 2 weeks. Their task will be collecting 10 virtual cubes one-by-one and putting them in the virtual treasure box. Clinical tests (Box and Blocks Test and motor part of the UPDRS) will be carried out in the clinical settings prior and after the training sessions. We hypothesise that the different feedback equipment may provide different results.

DETAILED DESCRIPTION:
The participants will practise grab and grasp in virtual environment (VE), either on a laptop computer or using 3D goggles. They will sit in a comfortable chair, with a small camera tracking the hand and finger movements of their affected (dominant, in case of both hands affected) hand. The participant will grab any of the virtual cubes lying around the VE and put it in the treasure box. When the cube falls into the treasure box it disappears and the participant scores, one by one until the 10th cube or 120s of time elapse. The cubes will be randomly spread in the VE and will all have the same virtual size, weight and bouncing factor, but different colour. If the participant is left-handed, the treasure box will be mirrored to the right side. If the cube is pushed into the floor, it disappears without a score and is lost. Each participant will take 10 consecutive training sessions in 2 weeks, each session lasting for 30min. Within a session, the participant will take 5 trials, with breaks of 1-2 min between them.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease diagnosis
* minor problems with daily activities and upper extremities
* Hoehn and Yahr Scale level 2-3

Exclusion Criteria:

* insufficient cognitive and motor abilities to carry out the exergaming task

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2018-12-16 (Actual); Study Completion 2018-12-16 (Actual)

PRIMARY OUTCOMES:
UDPRS III Motor | DIfference between the two assessments - a day or two before the first training sessions and immediately after the last training session
  Unified Parkinson's Disease Rating Scale Motor Function Part - difference score
BBT | DIfference between the two assessments - a day or two before the first training sessions and immediately after the last training session
  Box & Blocks Test - difference score

CONTACTS AND LOCATIONS:
Overall Officials: Imre Cikajlo, PhD, Principal Investigator — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cikajlo I, Peterlin Potisk K. Advantages of using 3D virtual reality based training in persons with Parkinson's disease: a parallel study. J Neuroeng Rehabil. 2019 Oct 17;16(1):119. doi: 10.1186/s12984-019-0601-1. PMID 31623622